CLINICAL TRIAL: NCT01074710
Title: A Phase I, Double-Blind, Placebo-Controlled, Randomized, 3-Period, Safety and Pharmacokinetic Study of 13C-uracil in a Semi-solid Meal at Single Oral Doses of 50, 100, and 200 mg in Healthy Volunteers
Brief Title: Safety and Pharmacokinetic Study of C13-URA in Healthy Volunteers
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Otsuka Pharmaceutical Co., Ltd. (Industry)
Responsible Party: Suguru Akamatsu/Director, R&D Department, Diagnostic Division
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Diagnostic
Other Study IDs: URA-09-001
Record Dates: First submitted 2010-02-18; First posted 2010-02-24 (Estimated); Last update posted 2010-07-19 (Estimated); Status verified 2010-05

CONDITIONS: Gastroparesis
MeSH Terms: conditions — Gastroparesis | interventions — Uracil

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- C13-URA (Experimental): administered C13-URA 50, 100, 200mg in same subjects
  Interventions: Drug: [2-13C] uracil
- Placebo (Placebo Comparator): 2 same subjects
  Interventions: Drug: [2-13C] uracil, placebo

INTERVENTIONS:
Drug: [2-13C] uracil — po, in the form of semi-solid meal, granules, once a period
  Arms: C13-URA
Drug: [2-13C] uracil, placebo — po, in the form of semi-solid meal, granules, once a period
  Arms: Placebo

SUMMARY:
The purpose of this study is to evaluate the safety and establish the pharmacokinetic (PK) profile of C13-URA in healthy volunteers

DETAILED DESCRIPTION:
The C13-URA Breath Test Kit is intended to be used as a diagnostic tool to identify rapid and/or delayed gastric emptying in patients who have upper GI symptoms such as stomach pain, fullness, early satiety, vomiting, etc., and who have suspected gastric emptying abnormalities such as gastroparesis or dumping syndrome.

This study will be a double-blind, placebo-controlled, 3-period safety and PK study of 13C-uracil administered as a single oral dose of 50 mg at step 1 (Period 1), 100 mg at step 2 (Period 2), and 200 mg at step 3 (Period 3) in the form of a semi-solid meal to subjects following at least a 10-hour fast from food and 2-hour fast from water. Dosing will be followed by a 6-hour fast from food and a 4-hour fast from water. There will be a washout of at least 7 days between doses.

The objectives of this study are as follows;

1)to evaluate the safety of 13C-uracil in a semi-solid meal in healthy volunteers, 2)to establish the pharmacokinetic profile of 13C-uracil in a semi-solid meal in healthy volunteers, 3)to assess the correlation between plasma concentration of 13C-uracil and urinary excretion of 13C-uracil, 4)to evaluate the reproducibility (intra/inter-individual variance) of the breath test, 5)to determine the dose for 13C-uracil that facilitates adequate Δ13C in breath expired by healthy volunteers

ELIGIBILITY:
Inclusion Criteria:

* Body mass index [range is 18.5 to 29.9 kg/m2]
* In good health, determined by no clinically significant findings from medical history, physical examination, 12-lead ECG, and vital signs

Exclusion Criteria:

* Significant history or clinical manifestation of any significant metabolic, allergic, dermatological, hepatic, renal, hematological, pulmonary, cardiovascular, gastrointestinal, neurological, or psychiatric disorder (as determined by the investigator)
* History of significant hypersensitivity, intolerance, or allergy to any drug compound, food, or other substance, unless approved by the investigator
* History of stomach or intestinal surgery or resection that would potentially alter absorption and/or excretion of orally administered drugs (except that appendectomy, hernia repair, and/or cholecystectomy will be allowed)
* History or presence of an abnormal ECG, which, in the investigator's opinion, is clinically significant

Ages: 18 Years to 50 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 8 (Actual)
Dates: Start 2010-02; Primary Completion 2010-05 (Actual); Study Completion 2010-05 (Actual)

PRIMARY OUTCOMES:
PK parameters | 6 hours
  Pharmacokinetic endpoints will include apparent clearance (CL/F), AUCt, AUC∞, Cmax, tmax, and t1/2,Z for 13C-uracil and its metabolites. The PK linearity and correlation between plasma concentration and urine excretion will be evaluated. Expired 13CO2 concentrations (Δ13C) will be converted to 13CO2-excretion(% dose/hr) to assess breath PK parameters (AUCt, AUC∞, Cmax, tmax, λZ, and t1/2,Z).

CONTACTS AND LOCATIONS:
Overall Officials: Stephen D Flach, MD, PhD, CPI, Principal Investigator — Covance Clinical Pharmacology, Inc.
Locations (1):
- Covance Clinical Pharmacology, Inc., Madison, Wisconsin, United States